CLINICAL TRIAL: NCT07401368
Title: Clinicians' Trust and Decision-Making Using AI-Based Fetal Growth Estimates With and Without Uncertainty: A Randomized Questionnaire Study
Brief Title: Clinicians' Trust in AI-Based Fetal Growth Estimates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Slagelse Hospital (Other); Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Zahra Bashir, Dr., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: F-25022462
Record Dates: First submitted 2026-01-23; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Fetal Growth; Obstetric Ultrasonography; Pregnancy; Clinical Decision-making
Keywords: Clinical decision-making; Artificial intelligence; Fetal weight estimation; Obstetric ultrasound; Trust; Human-AI interaction; Questionnaire study

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either an intervention group receiving information about AI model performance or a control group without such information. Groups are assessed in parallel.
Who Masked: Participant
Masking Description: Participants are unaware of their allocation to the control or intervention group and are not informed that different versions of the questionnaire exist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - No AI Performance Information (No Intervention): Participants complete the questionnaire without receiving information about the AI model's overall performance.
- ntervention - AI Performance Information (Other): Participants receive brief information about the AI model's overall performance before completing the questionnaire.
  Interventions: Other: Intervention - AI Performance Information

INTERVENTIONS:
Other: Intervention - AI Performance Information — Participants receive brief information about the AI model's overall performance before completing the questionnaire.
  Arms: ntervention - AI Performance Information

SUMMARY:
This study examines how clinicians trust and use artificial intelligence (AI) when estimating fetal weight during pregnancy.

Accurate assessment of fetal growth is important for identifying growth problems that may affect pregnancy management. New AI-based tools can estimate fetal weight from ultrasound images, but little is known about how clinicians trust these estimates or how uncertainty information influences their decisions.

In this study, clinicians will review anonymized ultrasound cases and compare fetal weight estimates generated by an AI model with traditional estimates. Some clinicians will also be shown information about the AI model's performance and uncertainty, while others will not.

Participants will be asked to choose which estimate they find most reliable, indicate their level of confidence, and decide whether they would recommend follow-up scans. The study aims to better understand how AI and uncertainty information affect clinical decision-making and trust among clinicians with different levels of experience.

DETAILED DESCRIPTION:
This is a randomized, matched, vignette-based questionnaire study designed to investigate clinicians' trust in and use of AI-based fetal growth estimates.

Clinicians from obstetrics and gynecology departments will be recruited and stratified by experience level. Participants will be randomized to either a control group or an intervention group. The intervention group will receive brief information about the AI model's overall performance, while the control group will not receive this information.

Each participant will assess a set of anonymized third-trimester ultrasound cases. For each case, clinicians will be presented with standard ultrasound images and relevant clinical context. They will be shown fetal weight estimates generated by an AI-based model and by a traditional biometric method, with or without accompanying uncertainty information in the form of confidence intervals.

For each case, clinicians will select the estimate they consider most clinically reliable, rate their confidence in that choice, and indicate whether they would recommend a follow-up growth scan. Case sets are matched by clinical experience, ensuring that identical cases are evaluated by clinicians with similar backgrounds across study arms.

The study focuses on clinicians as participants and involves no patient intervention. All ultrasound data are fully anonymized. The results will provide insight into how AI-generated estimates and uncertainty information influence clinical trust, preferences, and decision-making in fetal growth assessment.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians working in obstetrics and gynecology departments.
* Regular use of obstetric ultrasound in clinical practice.
* Willingness to participate in a questionnaire-based study.

Exclusion Criteria:

* Clinicians who do not perform obstetric ultrasound examinations.
* Clinicians with a known conflict of interest related to the AI system being evaluated.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinicians' choice of fetal weight estimation method | Immediately after questionnaire completion
  The proportion of cases in which clinicians choose the AI-based fetal weight estimate rather than the traditional Hadlock estimate when assessing anonymized ultrasound cases.

SECONDARY OUTCOMES:
Clinicians' confidence in selected fetal weight estimate | Immediately after questionnaire completion
  Clinicians' self-reported confidence in the selected fetal weight estimate, measured on a 7-point Likert scale for each case.
Recommendation of follow-up growth scan | Immediately after questionnaire completion
  Whether clinicians recommend a follow-up fetal growth scan based on the selected fetal weight estimate, recorded as a binary outcome (yes/no).
Impact of uncertainty information on model preference | Immediately after questionnaire completion
  Difference in clinicians' preference for AI-based versus traditional fetal weight estimates when AI predictions are presented with versus without uncertainty information.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Slagelse Hospital, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: No